CLINICAL TRIAL: NCT05758389
Title: A Prospective Single-center, Single-arm Clinical Study of the PD-1 Inhibitor Tislelizumab Combined With APF Sequential Surgery or Radical Concurrent Chemoradiotherapy in the Treatment of Locally Advanced Head and Neck Tumors
Brief Title: Tislelizumab Combined APF Chemotherapy in the Treatment of Locally Advanced Head and Neck Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Jing Yan, Deputy Director of the Department of Oncology, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-666-02
Record Dates: First submitted 2023-01-17; First posted 2023-03-07 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Head and Neck Tumors
Keywords: Immune checkpoint inhibitors; Chemotherapy; Locally advanced head and neck tumors; Induction therapy
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — tislelizumab; Paclitaxel; Cisplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- immunotherapy combined with chemotherapy (Experimental)
  Interventions: Drug: Tislelizumab, Paclitaxel (albumin-bound type), Cisplatin, 5-FU

INTERVENTIONS:
Drug: Tislelizumab, Paclitaxel (albumin-bound type), Cisplatin, 5-FU — evaluate the efficacy and safety of immunotherapy combined with chemotherapy

SUMMARY:
The goal of this clinical trial is to test in describe participant population. The main questions it aims to answer are:

1. evaluate the efficacy and safety of tislelizumab combined with APF sequential surgery or radical concurrent chemoradiotherapy in the treatment of locally advanced head and neck tumors.
2. the exploration of efficacy-related immune microenvironment genes Participants will receive tislelizumab combined with APF sequential surgery or radical concurrent chemoradiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old;
2. Histological or cytology-confirmed head and neck tumors (including oral, oropharynx, hypopharynx, larynx) squamous cell carcinoma, etc.;
3. Have at least one radiographically measurable lesion (RECIST 1.1 criteria);
4. The clinical stage is III-IVb (P16-) or II-III (P16+);
5. There are tumor samples that can detect gene expression;
6. ECOG score 0-1 points;
7. Have not received radiotherapy and chemotherapy or other anti-tumor drugs before;
8. The following hematological indicators need to be met: (1) Neutrophil count≥ 1.5×109/L; (2) Hemoglobin≥ 10g/dL; (3) Platelet count ≥ 100×109/L
9. The following biochemical indicators need to be met: (1) Total bilirubin ≤1.5× upper limit of normal value (ULN); (2) AST and ALT < 1.5 ×ULN; (3) Creatinine clearance ≥ 60ml/min; (4) Alkaline phosphatase ≤ 5 times ULN; (5) Activated partial thromboplastin time (APTT) and international normalized ratio (INR) ≤1.5xULN (for anticoagulation at a stable dose such as low molecular weight heparin or warfar.) LIN and INR can be screened within the expected therapeutic range of anticoagulants)
10. Subjects of childbearing age need to take appropriate protective measures (contraceptive measures) before enrollment and in trials administration or other methods of birth control);
11. Have signed informed consent;
12. Ability to follow study protocols and follow-up procedures.

Exclusion Criteria:

1. Received anti-tumor treatment in the past 6 months, including radiotherapy and chemotherapy, surgery, immunotherapy Wait;
2. Previously or concurrently suffering from other malignant tumors (except for malignant tumors that have been cured and survived for more than 5 years without cancer, such as skin basal cell carcinoma, cervical carcinoma in situ, superficial bladder cancer, and thyroid papillary carcinoma, etc.);
3. There is distant metastasis;
4. Active autoimmune diseases, history of autoimmune diseases (such as interstitial pneumonia, colitis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism, including but not limited to these diseases or syndromes); but excludes autoimmune-mediated hypothyroidism on stable doses of thyroid replacement hormone; type 1 diabetes on stable doses of insulin; vitiligo or resolved childhood asthma/allergies, Patients who do not require any intervention after adulthood;
5. Known history of primary immunodeficiency (including positive HIV test, or suffering from other acquired or congenital immunodeficiency diseases, or history of organ transplantation and allogeneic bone marrow transplantation);
6. Severe infection (CTC AE>2 grade) occurred within 4 weeks before the first use of the study drug, such as severe pneumonia requiring hospitalization, bacteremia, infection complications, etc.; baseline chest imaging examination showed active lung Inflammation, symptoms and signs of infection within 2 weeks before the first use of the study drug or the need for oral or intravenous antibiotic treatment (excluding prophylactic use of antibiotics);
7. The subject has severe liver and kidney dysfunction, HIV infection, HCV infection, uncontrolled clinical symptoms or diseases of the heart, such as: heart failure above NYHA grade II or echocardiography showing left ventricular ejection fraction (LVEF) < 50%; unstable angina; myocardial infarction within 1 year; patients with clinically significant supraventricular or ventricular arrhythmias requiring clinical intervention (including QTc interval ≥ 470 ms); uncontrolled diabetes, uncontrolled Patients with high blood pressure, hypertensive crisis or hypertensive encephalopathy or other diseases considered by the researchers to be ineligible;
8. Patients with untreated chronic hepatitis B or chronic hepatitis B virus (HBV) DNA exceeding 500 IU/ml, or patients with active hepatitis C virus (HCV) should be excluded; inactive hepatitis B surface Antigen carriers, treated and stable hepatitis B patients (HBV DNA<500IU/ml), and cured hepatitis C patients can be enrolled;
9. Have a history of interstitial lung disease (excluding radiation pneumonitis that has not been treated with hormones) and non-infectious pneumonia;
10. Active tuberculosis infection was found through medical history or CT examination, or patients with a history of active tuberculosis infection within 1 year before enrollment, or patients with a history of active tuberculosis infection more than 1 year ago but without formal treatment;
11. Patients who have received any of the following treatments (1) Subjects who need to be given corticosteroids (> 10 mg prednisone equivalent dose per day) or other immunosuppressants for systemic treatment within 2 weeks before the first use of the study drug, except for local inflammation and prevention of allergies and nausea, Cases of use of corticosteroids for vomiting. In the absence of active autoimmune disease, corticosteroid replacement with inhaled or topical steroids and curative doses of prednisone >10 mg/day is permitted; (2) Have been vaccinated against tumors; those who have been vaccinated or have been vaccinated with live vaccines within 4 weeks before the first administration of the study drug; (3) Received major surgery or severe trauma within 4 weeks before the first use of the study drug; (4) Enrolled in another clinical study at the same time;
12. Pregnant and lactating women. Women of childbearing age must take a pregnancy test within 7 days before enrollment Negative;
13. Substance abuse, clinical or psychological or social factors that hinder informed consent or research conduct influences;
14. Those who may be allergic to the study drug;
15. Those who cannot perform radiotherapy and chemotherapy due to social or geographical factors;
16. Significant weight loss within 6 weeks before enrollment (weight loss ≥ 10%);
17. Any uncertain factors affecting the safety or compliance of the subjects;
18. Contraindications to hormone use.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-08-07 (Actual); Study Completion 2025-12-07 (Estimated)

PRIMARY OUTCOMES:
Change of pathological examination | Change from Baseline pathologic examination at the end of Cycle 3 (each cycle is 21 days)
  Changes in pathologic examination before treatment and after 3-cycle induction therapy were evaluated to derive the number and proportion of patients with pathological complete remission
Change of tumor size | Change from baseline tumor size at the end of Cycle 3 (each cycle is 21 days)
  imaging (MRI or CT) assessment according to RECIST v1.1 was performed and documented during follow-up as required

SECONDARY OUTCOMES:
Security assessment | At the end of Cycle 3 (each cycle is 21 days)
  according to the NCI-CTCAE 4.0 adverse reaction evaluation criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Oncology, Drum Tower Hospital, Nanjing University School of Medicine, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided